CLINICAL TRIAL: NCT06604884
Title: Neurovascular Product Surveillance Registry (NV PSR INSPIRE) Pipeline™ Vantage Embolization Device With Shield Technology™ Post Approval Study (PAS)
Brief Title: NV PSR INSPIRE-A Pipeline™ Vantage Post Approval Study
Status: Recruiting | Type: Observational
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT24028
Record Dates: First submitted 2024-09-17; First posted 2024-09-20 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Treatment of Intracranial Aneurysms — Embolization of aneurysms using the Pipeline™ Vantage Embolization Device with Shield Technology™

SUMMARY:
The purpose of the Pipeline™ Vantage Embolization Device with Shield Technology™ Post Approval Study (PAS) ("Pipeline™ Vantage PAS") is to collect safety and effectiveness data in patients undergoing treatment for intracranial aneurysms (IA) using the Pipeline™ Vantage Embolization Device with Shield Technology™ ("Pipeline™ Vantage Device") in a post approval setting.

DETAILED DESCRIPTION:
The INSPIRE Pipeline™ Vantage Post Approval Study is a, prospective, multi-center, single-arm clinical study to collect safety and effectiveness data in patients undergoing treatment for intracranial aneurysms using the Pipeline™ Vantage Embolization Device with Shield Technology™.

This study is a sub-study to the Neurovascular Product Surveillance Registry (NCT02988128).

ELIGIBILITY:
Inclusion Criteria:

1. Patient or legally authorized representative (LAR) has provided written informed consent using the Ethics Board and Medtronic approved Informed Consent Form and agrees to comply with the protocol requirements. HIPAA/data protection authorization has been provided and signed by the patient (or patient's LAR) as applicable per local law.
2. Patient has an intracranial aneurysm intended to be treated with the Pipeline™ Vantage Embolization Device with Shield Technology™.
3. Patient is an adult per local law at time of consent.

Exclusion Criteria:

1. Patient with any contraindications for the device or procedure per the Pipeline™ Vantage Device local geography IFU.
2. Patient who may be unable to complete the study follow-up.
3. The Investigator determined that the health of the patient may be compromised by the patient's enrollment.
4. Female patient who is known to be pregnant or is breastfeeding or wishes to become pregnant during participation in the study.
5. Patient is currently enrolled in, or plans to enroll in, any concurrent drug/device study that may confound the study results.

Min Age: 22 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients requiring treatment for intracranial aneurysms with the market approved Pipeline™ Vantage Embolization Device with Shield Technology™ device are eligible for the registry
Sampling Method: Non-Probability Sample
Enrollment: 118 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2033-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of the composite outcome (Occlusion of the target aneurysm, Significant parent artery stenosis, Retreatment of the target aneurysm) at 1 year post-procedure. | 1 Year
  Incidence of complete occlusion of the target intracranial aneurysm (Raymond-Roy I) without significant parent artery stenosis (≤ 50%) nor re-treatment of the target intracranial aneurysm at 1-year post-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Harsh Sancheti, Study Director — Medtronic
Locations (2):
- United States (2):
  - Wellstar Research Institute, Marietta, Georgia
  - McLaren Healthcare, Flint, Michigan

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be available